CLINICAL TRIAL: NCT03923660
Title: Ventilatory Adaptation to Concentric Versus Eccentric Exercise in Patients With Severe COPD
Acronym: CONvEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P/2018/374
Record Dates: First submitted 2019-04-02; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2018-09

CONDITIONS: Chronic Obstructive Pulmonary Disease Severe
Keywords: COPD; breathing pattern; exercise; concentric; eccentric
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concentric-eccentric (Experimental): Concentric-eccentric
  Interventions: Other: Incremental Concentric-eccentric exercise test
- Eccentric-concentric (Experimental): Eccentric-concentric
  Interventions: Other: Incremental Eccentric-concentric exercise test

INTERVENTIONS:
Other: Incremental Concentric-eccentric exercise test — Patients will perform incremental exercise test on semi recumbent eccentric ergometer
  Arms: Concentric-eccentric
Other: Incremental Eccentric-concentric exercise test — Patients will perform incremental exercise test on semi recumbent concentric ergometer
  Arms: Eccentric-concentric

SUMMARY:
Pulmonary rehabilitation (PR) based on concentric exercise training has become an integral component in the treatment of patients with chronic obstructive pulmonary disease (COPD), improving functional capacities while diminishing symptoms and improving quality of life.

However, the response to concentric exercise training is heterogeneous from one COPD patient to another. The inability of some COPD patients to achieve the exercise intensities required to stress limb muscles due to severe ventilatory limitation could partially explain their poor response to training.

Endurance exercise with eccentric muscle contractions could be an interesting alternative to concentric exercise because it produces greater muscle force through its lower metabolic cost. Eccentric exercise could allow patients with severe airflow limitation to perform prolonged exercise sessions with sufficient intensity to improve muscle function.

Nevertheless, a recent study performed in healthy young subjects reported that eccentric exercise induced a more hyperpneic breathing pattern (i.e., lower tidal volume and higher breathing frequency) that concentric for a given minute ventilation.

The main objective of CONvEX study is to compare ventilatory adaptation between two modalities of exercise performed on cycle ergometer (concentric versus eccentric) in severe COPD patients.

DETAILED DESCRIPTION:
Pulmonary rehabilitation (PR) based on concentric exercise training has become an integral component in the treatment of patients with chronic obstructive pulmonary disease (COPD), improving functional capacities while diminishing symptoms and improving quality of life.

However, the response to concentric exercise training is heterogeneous from one COPD patient to another. The inability of some COPD patients to achieve the exercise intensities required to stress limb muscles due to severe ventilatory limitation could partially explain their poor response to training.

Endurance exercise with eccentric muscle contractions could be an interesting alternative to concentric exercise because it produces greater muscle force through its lower metabolic cost. Eccentric exercise could allow patients with severe airflow limitation to perform prolonged exercise sessions with sufficient intensity to improve muscle function.

Nevertheless, a recent study performed in healthy young subjects reported that eccentric exercise induced a more hyperpneic breathing pattern (i.e., lower tidal volume and higher breathing frequency) that concentric for a given minute ventilation.

The main objective of CONvEX study is to compare ventilatory adaptation between two modalities of exercise performed on cycle ergometer (concentric versus eccentric) in severe COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Severe COPD (FEV1 [forced expiratory volume in 1 second] / FVC [forced vital capacity] < 70% et FEV1 < 50%)
* Informed consent
* Affiliation to a social security scheme

Exclusion Criteria:

* Effort oxygen therapy
* Cardiovascular, neuromuscular or musculoskeletal disorders that can provide significant dyspnea or limit exercise
* Legal incapacity
* Low or no cooperation anticipated

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Ventilatory adaptation | week 1
  Breathing frequency/tidal volume ratio at the maximum common minute ventilation.

SECONDARY OUTCOMES:
Dynamic hyperinflation | week 1
  Dynamic hyperinflation will be assessed through iterative inspiratory capacity (IC) measurment during exercise. A decrease in IC >150 mL compared to resting levels at any time point during exercise will be considered as dynamic hyperinflation.
Brachial muscle enrollment | week 1
  2.4 GHz electromyographic activity of biceps brachii recorded using surface electrod (Cometa Wave Plus wireless EMG)
Quadriceps muscle enrollment | week 1
  2.4 GHz electromyographic activity of vastus lateralis recorded using surface electrod (Cometa Wave Plus wireless EMG)
Ventilatory efficiency | week 1
  Dead volume/Tidal volume ratio
Ventilatory efficiency | week 1
  Minute ventilation/Carbon dioxide production ratio
Tolerance | week 1
  Borg modified scale [ranging from 0 to 10] for dyspnoea 0 indicates no dyspnoea and 10 the maximum dyspnoea

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France